CLINICAL TRIAL: NCT02425592
Title: Active Surveillance in Prostate Cancer, Imaging to Detect Radiographic Progression as an Endpoint (ASPIRE)
Acronym: ASPIRE
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1501015246
Record Dates: First submitted 2015-04-16; First posted 2015-04-24 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Men on Active Surveillance: This study will include men between age 30-80 with Gleason 6 prostate cancer, prostate specific antigen (PSA) <20, clinical stage <cT3, and a life expectancy of at least ten years. To be eligible, men must have undergone an MRI-USG fusion prostate biopsy for an elevated PSA or abnormal prostate examination that demonstrates Gleason 6 prostate cancer. If a man is already on active surveillance, the MRI-USG fusion biopsy may be negative or confirm Gleason 6 prostate cancer. Eligible men will be approached at their post fusion-biopsy visit to discuss the biopsy results and offered enrollment in the trial.

SUMMARY:
The objective in this study is to determine if MRI-identified progression can decrease frequency or need for repeated prostate biopsy in men on active surveillance (AS).

Our hypothesis is that MRI alone is adequate to detect progression of prostate cancer in men on active surveillance (AS) after a MRI-US fusion prostate biopsy.

DETAILED DESCRIPTION:
MRI Fusion prostate biopsy will transform Active Surveillance (AS) for men with low risk prostate cancer. Treatment for prostate cancer, usually surgical removal or radiation delivered to the whole prostate, is associated with significant morbidity including incontinence and impotence.

The goal of this and future research is to maximize the effectiveness of prostate imaging in order to minimize the morbidity of prostate biopsy and hence improve the quality of life of patients with prostate cancer. There are many applications to improved imaging of prostate cancer, but several the investigators are interested in include: improved risk stratification to limit unnecessary treatment while providing appropriate treatment to prevent progression; limiting the number of biopsies needed for diagnosis and/or decreasing the frequency of biopsies and hence decreasing biopsy-related morbidity; focal therapy for confirmed focal disease rather than treating the entire prostate in order to limit the significant morbidity associated with whole-gland treatment.

This is an investigator-initiated, multi-center, prospective observational phase II trial evaluating MRI to detect prostate cancer progression in patients with low risk prostate cancer on Active Surveillance. The two centers involved will be the Yale-New Haven Hospital Smilow Cancer Center (Yale) and the VA Connecticut Healthcare System (VACT). The Yale School of Medicine will serve as the central data-coordinating center for this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80
* Completed MRI Fusion prostate biopsy either in the past that demonstrated Gleason 6 prostate cancer and are either currently enrolled in Active Surveillance or are interested in Active surveillance, or have completed an MRI Fusion prostate biopsy at the first visit that demonstrates Gleason 6 prostate cancer and are interested in Active Surveillance
* Diagnosed with Gleason 6 prostate cancer
* PSA <20
* <cT3 prostate cancer
* Ability to receive an MRI with IV gadolinium contrast
* Life expectancy >10 years (by physician estimate)
* Understanding and willingness to provide consent
* English speaking

Exclusion Criteria:

* Received treatment for prostate cancer (hormone manipulation, surgery, radiation).
* Known metastatic disease
* High risk prostate cancer by Epstein Criteria
* Any Gleason 7 or higher prostate cancer on prostate biopsy
* Inability to receive an MRI with IV gadolinium contrast
* Life expectancy <10 years
* Unwillingness to undergo monitoring and imaging studies
* Non-English speaking

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include men between age 30-80 with Gleason 6 prostate cancer, PSA <20, <cT3, and a life expectancy of at least ten years.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2025-05 (Actual)

PRIMARY OUTCOMES:
Tumor Histologic Progression Rate | 3 years
  MRI-US Fusion biopsy
Tumor Radiologic Progression Rate | 3 years
  MRI

SECONDARY OUTCOMES:
Anxiety Using Cancer Distress Thermometer Scores | 3 years
  serial anxiety measurements on standardized scale
Urinary Function Using International Prostate Symptom Scores | 3 years
  monitoring urinary symptoms using standardized questionnaire
Erectile Function Using Sexual Health Inventory for Men Scores | 3 years
  monitoring sexual function as measured by standardized questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Preston Sprenkle, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - VA Connecticut Healthcare System (VACT), West Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No